CLINICAL TRIAL: NCT07271537
Title: Outcomes of Karydakis Versus Limberg Flap for the Management of Primary Sacrococcygeal Pilonidal Sinus
Brief Title: Karydakis Versus Limberg Flap for the Management of Primary Sacrococcygeal Pilonidal Sinus
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, professour, Zagazig University
Other Study IDs: pilonidal sinus
Record Dates: First submitted 2025-11-13; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Pilonidal Cyst and Sinus Without Abscess
Keywords: pilonidal sinus; karydakis; limberg flap
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Karadakis flap: Karadakis flap for managing pilonidal cyst
  Interventions: Procedure: karydakis surgery
- Limberg flap
  Interventions: Procedure: Limberg flap

INTERVENTIONS:
Procedure: karydakis surgery — karydakis surgery for managing pilonidal sinus
  Groups: Karadakis flap
Procedure: Limberg flap — using rheumboid flap to cover the defect after pilonidal sinus excision
  Groups: Limberg flap

SUMMARY:
study comparing the Karydakis and Limberg flaps

DETAILED DESCRIPTION:
study comparing the Karydakis and Limberg flaps in management of pilonidal sinus

ELIGIBILITY:
Inclusion Criteria:

* sexually active,
* employed or driving ,
* patients diagnosed with sacrococcygeal primary symptomatic pilonidal sinus based on clinical aspects, physical examination, and disease-specific history

Exclusion Criteria:

* lost follow up
* refuse surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients > 18 years with PNS underwent karydakis and limberg flap
Sampling Method: Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
sexual function comparison | 1 year
  sexual function evaluation through questionnaire modulated by our group and asked to the patients

SECONDARY OUTCOMES:
driving function evaluation | 1 year
  driving evaluation after surgery through questionnaire modulated by our group and asked to the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable requirement
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Oetzmann von Sochaczewski C, Godeke J. Pilonidal sinus disease on the rise: a one-third incidence increase in inpatients in 13 years with substantial regional variation in Germany. Int J Colorectal Dis. 2021 Oct;36(10):2135-2145. doi: 10.1007/s00384-021-03944-4. Epub 2021 May 16. PMID 33993341